CLINICAL TRIAL: NCT05536154
Title: Prospective, Single-arm, Multicenter Exploratory Clinical Study of the Combination of Etoposide, Cytarabine and PEG-rhG-CSF (EAP Regimen) as First Line Mobilization Regimen of Hematopoietic Stem Cells in Patients With Hematological Malignancies
Brief Title: Etoposide+Cytarabine+PEG-rhG-CSF as First Line Mobilization Regimen of Hematopoietic Stem Cells in Patients With Hematological Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated People's Hospital of Ningbo University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-YAN-030
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Lymphoma; Multiple Myeloma
Keywords: Etoposide; Cytarabine; PEG-rhG-CSF; Hematological Malignancies; Hematopoietic Stem Cell Mobilization
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Hematologic Neoplasms | interventions — Etoposide; Cytarabine; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EAP regimen (Experimental): The combination regimen of etoposide, cytarabine and PEG-rhG-CSF.
  Interventions: Drug: Etoposide; Drug: Cytarabine; Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: Etoposide — Day 1~Day 2: 75mg/m^2
  Other Names: VP-16
Drug: Cytarabine — Day 1~Day 2: 200mg/m^2, q12h
  Other Names: Ara-C
Drug: PEG-rhG-CSF — Day 6: 6mg

SUMMARY:
This is a single-arm, multicenter, exploratory clinical study to evaluate the safety and efficacy of the combination of etoposide, cytarabine and PEG-rhG-CSF (EAP regimen) as first line mobilization regimen of hematopoietic stem cells in patients with lymphoma and multiple myeloma. All eligible patients will receive EAP regimen treatment, then the number of CD34+ cells and white blood cells will be monitoring. When the collection standard is met, hematopoietic stem cell collection will be started.

DETAILED DESCRIPTION:
In patients older than 65 years, or with creatinine >2.5 mg/dL but with an endogenous creatinine clearance >50%, the dose of etoposide and Ara-C should be reduced by one-quarter to one-third.

Routinely blood analyses and peripheral blood CD34+ cells monitored will be performed daily from day 9 to the end of HSC collection or the abandonment of HSC collection. If the WBC count is ≤10×109/L, 5μg/kg/d of G-CSF should be injected subcutaneously until the end of HSC collection.

Leukapheresis can be performed when the white blood cell counts recover (WBC count was≥4×109/L) following chemotherapy and the CD34+ cell count was≥20/μL. Leukapheresis started if the peripheral blood CD34+ counts plateaued at ≥5 cells/μL and <20 cells/μL after recovery of white blood cell counts following chemotherapy, the clinician decided whether to add plerixafor based on the specific situation of the patient. Leukapheresis should be abandoned if the peak circulating CD34+ cells were <5/μL up to 20 days after chemotherapy. CD34+ cells were determined by multi-parameter flow cytometry and a dual-platform approach. Two blood cell separators were used at the study sites: Spectra-Optia Apheresis system (Terumo BCT, Lake-wood, CO, USA) , COM.TEC (Fresenius Kabi). During each leukapheresis, 2.5 times the patients' blood volume (±25%) had to be processed within 5 h.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as lymphoma or multiple myeloma, with auto-HSCT indication.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0~2.
3. Life expectancy ≥ 3 months.
4. Subjects must be able to understand the protocol and be willing to enroll the study, sign the informed consent, and be able to comply with the study and follow-up procedures.

Exclusion Criteria:

1. Patients with severe cardiac, hepatic or renal insufficiency, such as:

   * Serum direct bilirubin (DBIL)>2× upper limit of normal (ULN);
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2× ULN;
   * Serum creatinine clearance rate≤50%;
   * Cardiac function class II or higher or severe arrhythmia.
2. History of hematopoietic stem cell mobilization.
3. Patients with active infection.
4. Female subjects who are pregnant or lactating.
5. Subjects with any life-threatening disease, medical condition or organ system dysfunction compromising their safety or causing unnecessary risks for the study results in the investigator' opinion, such as unstable heart disease, stroke, rheumatoid arthritis, lupus.
6. Have received live vaccine and attenuated live vaccine within 4 weeks before enrollment.
7. History of allergy to Etoposide (VP-16), Cytarabine (Ara-C), or PEG-rhG-CSF.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
% of patients achieving the collection of ≥2×10^6 CD34+ cells/kg. | 4 weeks
  The proportion of patients whose cells can be successfully mobilized and collected with a target CD34+ Hematopoietic Stem Cell (HSC) dose of ≥2×10^6/kg.

SECONDARY OUTCOMES:
% of patients achieving the collection of #5×10^6 CD34+ cells/kg. | 4 weeks
  The proportion of patients whose cells can be successfully mobilized and collected with a target CD34+ Hematopoietic Stem Cell (HSC) dose of >5×10^6/kg.
TRAEs | 4 weeks
  Incidence and severity of treatment related adverse events (TRAEs). Adverse events will be collected based on NCI CTCAE version 5.0.
Time from PEG-rhG-CSF mobilization to HSC collection. | 4 weeks
  To determine the time period from PEG-rhG-CSF mobilization to successfully collection of HSC.
The average collection times of EAP scheme | 4 weeks
Hematopoietic reconstitution and therapeutic adverse events after transplantation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lu, Principal Investigator — The Affiliated People's Hospital of Ningbo University
Locations (14):
- China (14):
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou central hospital, Huzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Jinhua People's Hospital, Jinhua, Zhejiang
  - Lishui Municipal Central Hospital, Lishui, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing Hospital of Zhejiang University, Shaoxing, Zhejiang
  - Shaoxing Second Hospital, Shaoxing, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - The 2nd School of Medicine,WMU/The 2nd Affiliated Hospital and Yuying Children's Hospital of WMU, Wenzhou, Zhejiang